CLINICAL TRIAL: NCT06465134
Title: Mechanisms for Incident and Recurrent Atrial Fibrillation in Patients With Obstructive Sleep Apnea; AF - Milano Trieste Stockholm
Brief Title: Mechanisms for Atrial Fibrillation in Obstructive Sleep Apnea
Acronym: AF-MiTriSto
Status: Recruiting | Type: Observational
Sponsor: Danderyd Hospital (Other)
Collaborators: Istituto Auxologico Italiano (Other); University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: KAROLINSKA INSTITUTE, DANDERYD
Record Dates: First submitted 2024-03-26; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea; Hypertension; Autonomic Dysfunction; Arterial Stiffness
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Hypertension; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients scheduled for AF ablation or cardioversion
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
Atrial fibrillation (AF) is the most common rhythm disorder and involves an increased risk of cardiovascular disease and death, impaired quality of life and a high proportion of healthcare consumption. An important risk factor is obstructive sleep apnea (OSA). However, it is not fully understood why OSA induces AF. It may be due to a proinflammatory state, sympathetic activation and acute changes in blood pressure during apnéas, but few studies are performed. Hypertension with its coherent arterial stiffness is related to all these factors, is common in OSA, and is the most common cause of AF. The cause of AF in hypertensive subjects is believed due to a pressure overloaded left heart, with dilation and fibrosis of the left atrium, promoting the development of AF. Hypertension and arterial stiffness can thus be important triggering factors for AF in OSA.

In this project, teh investigators investigate the occurrence of OSA in AF patients. Furthermore, underlying mechanisms for the development and recurrence of AF after intervention in OSA patients are investigated.

300 patients scheduled for AF ablation or cardioversion are invited and examined with sleep registration, 24h blood pressure, aortic stiffness measurement, test of autonomic function, echocardiography, ECG and labs. The patients are followed at months 3, 6 and 12 with 7 days ECG for recurrence. The aim is to give insights into the need for screening for OSA in patients with AF. The study also aim at enabling preventive treatment through better understanding of underlying treatable mechanisms. The results are believed to lead to fewer new AFs, as well as fewer AF recurrences in patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years scheduled for AF ablation or cardioversion

Exclusion Criteria:

diagnosis of AF for more than 7 years

* previous cardiac surgery including AF ablation
* severe valvular heart disease
* diagnosed structural heart disease
* systolic function in sinus rhythm <50%.
* severe hypertensive heart disease or known hypertrophic heart disease (amyloidosis, hereditary hypertrophic heart disease)
* invalidating chronic diseases imaging material on echocardiography not of sufficient quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at San Luca Hospital Cattinara Hospital Italy, and Danderyd Hospital Sweden are used. Patients with atrial fibrillation scheduled for AF ablation or cardioversion are selected.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time to recurrence of AF measured on 7 days electrocardiography at month 3, 6, 12 | one year
  Recurrence of atrial fibrillation after AF ablation or cardioversion

SECONDARY OUTCOMES:
aortic stiffness measured by tonometry; pulse wave velocity (m/s) | baseline measurements
  measured aortic stiffness (measured as pulse wave velocity in m/s) in subjects with OSA compared to those without OSA in the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Lundwall, MD PhD, Principal Investigator — KAROLINSKA INSTITUTE, DANDERYD HOSPITAL; Gianfranco Parati, Professor, Principal Investigator — Istituto Auxologico Italiano
Locations (3):
- Italy (2):
  - San Luca Hospital, Milan
  - Cattinara Hospital, Trieste
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided